CLINICAL TRIAL: NCT00994409
Title: Berliner Schlaganfallregister - Nachbefragung Von Patienten Mit Schlaganfall
Brief Title: Patient Satisfaction in Stroke Patients
Acronym: PatZuFrie
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Center for Stroke Research Berlin (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Christian H Nolte MD, Dept. Neurology, Charite Campus Benjamin Franklin
Other Study IDs: CSB-PatZuFrie; EA4/019/08
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Stroke
Keywords: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this trial is to guarantee a follow-up of all stroke and transient ischemic attack (TIA) patients. With this follow-up assessment long term effects of therapy and prevention measures can be detected and monitored. It is part of quality assurance.

DETAILED DESCRIPTION:
Primary efficacy endpoint: Number of patients who state that they received all the information they want about the causes and nature of their illness Key secondary endpoint(s): Compliance/adherence with discharge medication. Re-events. Degree of Disability. Activities of daily living. Mortality.

ELIGIBILITY:
Inclusion Criteria:

* all patients eligible

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke and TIA patients treated at the Charite with acute stroke or TIA onset less than 7 days
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-07 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Primary efficacy endpoint: Number of patients who state that they received all the information they want about the causes and nature of their illness. | September 2010

SECONDARY OUTCOMES:
Compliance/adherence with discharge medication Activities of daily living | September 2010
Re-events | September 2010
Degree of Disability | September 2010
Mortality | September 2010

CONTACTS AND LOCATIONS:
Overall Officials: Peter U Heuschmann, Professor, Principal Investigator — Center for Stroke Research Berlin
Locations (1):
- Dept. Neurology, Charité Campus Benjamin Franklin, Berlin, Germany